CLINICAL TRIAL: NCT02652130
Title: Safety Follow-up Through 180 Days of Treatment With Remestemcel-L in Study MSB-GVHD001 in Pediatric Patients Who Have Failed to Respond to Steroid Treatment for Acute GVHD
Brief Title: Safety Follow-up of Treatment With Remestemcel-L in Pediatric Participants Who Have Failed to Respond to Steroid Treatment for Acute GVHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MSB-GVHD002
Record Dates: First submitted 2015-11-03; First posted 2016-01-11 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Grade B Acute Graft Versus Host Disease; Grade C Acute Graft Versus Host Disease; Grade D Acute Graft Versus Host Disease
Keywords: GVHD
MeSH Terms: interventions — remestemcel-l

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Safety population (Experimental): All participants who were enrolled and had received at least 1 dose of remestemcel-L in Study MSB-GVHD001.
  Interventions: Biological: Remestemcel-L

INTERVENTIONS:
Biological: Remestemcel-L — No intervention was given in Study MSB-GVHD002 (NCT02652130). It was a safety follow-up trial of remestemcel-L-treated participants from Study MSB-GVHD001.

SUMMARY:
Ongoing safety assessment follow-up to Protocol MSB-GVHD001 (NCT02336230) of remestemcel-L treatment in pediatric participants with acute graft versus host disease (aGVHD), following allogeneic hematopoietic stem cell transplant (HSCT), that have failed to respond to treatment with systemic corticosteroid therapy.

DETAILED DESCRIPTION:
This is a safety follow-up study through 180 days of remestemcel-L treatment in participants who took part in MSB-GVHD001. This study will also explore duration of response over time. Participants who took part in in MSB-GVHD001 and received at least one dose of remestemcel-L as outlined in that protocol will be evaluated at baseline (Day 100) and at Days 120, 140, 160 and 180 for safety endpoints. Participants who took part in Protocol MSB-GVHD001 and received the first 8 doses of remestemcel-L as outlined in that protocol will be evaluated at baseline (Day 100) and at Days 120, 140, 160 and 180 after initial remestemcel-L infusion for evidence of duration of response over time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have participated in MSB-GVHD001 and have received at least one infusion of remestemcel-L.
* Participant or participant's authorized representative must be capable of providing written informed consent. Assent, if applicable, must also be collected when required by the Institutional Review Board (IRB)/Ethics Committee (EC).
* Female participants of childbearing potential (≥ 10 years of age) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for the follow-up time period. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
* The participant must be willing and able to comply with study procedures, remain at the clinic as required during the study period, and return to the clinic for the follow-up evaluation as specified in this protocol.

Exclusion Criteria:

* The investigator believes it to be in the best interest of the participant not to participate in the safety follow-up study.
* Participant has participated or is currently participating in any autologous or allogeneic stem cell or gene therapy study for the treatment of aGVHD. Participants participating in investigative protocols aimed at modification of the transplant graft (such as T cell depletion) or aimed at modification of the conditioning regimen will be allowed in the study.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher James, Study Director — Mesoblast, Inc.
Locations (20):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - CHOC Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado Center for Cancer/Blood Disorders, Aurora, Colorado
  - Alfred I. duPont Hospital for Children of the Nemours Foundation, Wilmington, Delaware
  - Miami Children's Research Institute, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Children's Hospital at Montefiore, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 participants enrolled in Study MSB-GVHD001 [NCT02336230], received >=1 dose of remestemcel-L; evaluated up to Day100. These participants were followed-up for OS, GVHD activity up to Day180 (end of Study MSB-GVHD002 [NCT02652130]). 32 of 54 participants were enrolled in Study MSB-GVHD002; evaluated at Baseline (Day 100) and at Days120, 140, 160 and 180.
Groups:
- Remestemcel-L: All participants who were enrolled and had received at least 1 dose of remestemcel-L in Study MSB-GVHD001.
Period: Overall Study
Arm/Group | Remestemcel-L
Started | 32
Completed | 31
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who signed the informed consent form and received at least one dose of study treatment (complete or partial) in the study MSB-GVHD001 and who signed the informed consent form for the study MSB-GVHD002 were followed across both the studies MSB-GVHD001 and MSB-GVHD002.
Arm/Group | Remestemcel-L
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (5.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 20
  Race: Black or African American | 3
  Race: Asian | 2
  Race: American Indian or Alaska Native | 1
  Race: Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate Through Day 180
Description: The overall survival rate is defined as the percentage of participants alive at the given time point. OS is defined as the time to death from the start of drug therapy.
Time Frame: From Baseline Day 1 in the Study MSB-GVHD001 up to Day 180 in Study MSB-GVHD002 (180 days)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Remestemcel-L
Number analyzed (Participants) | 54
percentage of participants | 68.5

2. Secondary Outcome: Overall Survival Rate at Day 180 for Participants Who Had Overall Response (OR) at Day 28 of Study MSB-GVHD001
Description: as for outcome 1
Time Frame: From Baseline (Day 1) in the Study MSB-GVHD001 up to Day 180 in the Study MSB-GVHD002 (180 days)
Population: Duration of Response population included all participants who participated in Study MSB-GVHD001 and showed OR or very good partial response (VGPR) to remestemcel-L at Day 28 in Study MSB-GVHD001. The OS was evaluated across both Studies MSB-GVHD001 and MSB-GVHD002.
Measure: Number; unit: percentage of participants
Arm/Group | Remestemcel-L
Number analyzed (Participants) | 38
percentage of participants | 78.9

ADVERSE EVENTS:
Time Frame: Baseline (Day 100) up to Day 180 in Study MSB-GVHD002
Description: Safety population included all participants who signed the informed consent form and received at least one dose of study treatment (complete or partial) in Study MSB-GVHD001 and who signed the informed consent form for Study MSB-GVHD002. As no treatment was administered in this study, only serious adverse events are reported. Any non-serious treatment-emergent adverse events that occurred within 30 days of last treatment at the 5% threshold will be reported in Study MSB-GVHD001 [NCT02336230].
Arm/Group | Remestemcel-L
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 15/32
Other Adverse Events (participants affected / at risk) | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remestemcel-L (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 1
Nocardiosis (Infections and infestations) | 1
Osteomyelitis acute (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications (abstracts, posters or presentations) must be presented to the Publication Steering Committee for review prior to submission or public display and are not allowed prior to the publication of the primary manuscript, or eighteen (18) months from the conclusion of the Study. PI shall provide Sponsor a copy of any proposed public disclosure at least 30 days prior to submission. Sponsor may ask PI to delay the disclosure for a maximum of 60 days to file proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT02652130/Prot_SAP_000.pdf